CLINICAL TRIAL: NCT00791401
Title: The Pharmacokinetics of ER OROS Paliperidone in Subjects With Varying Degrees of Impaired Renal Function (Mild, Moderate, and Severe) as Compared to Subjects With Normal Renal Function
Brief Title: A Study of the Pharmacokinetics of ER OROS Paliperidone in Volunteers With Normal or Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004207
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia; Renal Impairment
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs; ER OROS Paliperidone
MeSH Terms: conditions — Schizophrenia; Renal Insufficiency; Mood Disorders

INTERVENTIONS:
Drug: ER OROS Paliperidone

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single oral dose of 3 mg extended release paliperidone (ER OROSÃ' paliperidone) in patients with varying degrees of renal impairment (mild, moderate, and severe), compared to patients with normal renal function. Secondary objectives include the assessing the disposition of the (+) and (-) enantiomers by means of an enantioselective liquid chromatography mass spectrometry assay, to determine plasma protein binding of the enantiomers in patients with impaired renal function, compared with patients with normal renal function, and to evaluate the tolerability and safety profile of ER OROS paliperidone in patients with varying degrees of renal impairment (mild, moderate, and severe) compared with patients with normal renal function.

DETAILED DESCRIPTION:
This is a single dose, parallel group, open-label, 2 center pharmacokinetic study, consisting of a pretreatment (screening) period of between 1 and 3 weeks, an open label treatment period (single dose of ER OROS paliperidone on Day 1 only, and with end of study procedures and discharge ending on Day 6). All patients will be screened between Day 21 and Day 1 for renal function. On Day 1, all patients will receive a single oral dose of 3 mg ER OROS paliperidone and undergo a 120 hour follow up with serial blood collections for pharmacokinetics, safety and tolerability assessments. Patients will be discharged after giving a pharmacokinetic blood sample and completing end of study assessments in the morning of Day 6. Group matching will be applied to the renal function groups to reduce bias and increase comparability of age, weight, gender, and ethnicity. This study is aimed to compare the pharmacokinetics and safety profile of ER OROS paliperidone in patients with varying degrees of renal impairment with that of normal patients. 3 mg oral ER OROS paliperidone

ELIGIBILITY:
Inclusion Criteria:

* All patients: A body mass index (weight [kg]/height (m)²) in the range of 18.0 to 32.0 kg/m², inclusive
* Patients with normal renal function: Healthy on the basis of a prestudy physical examination, medical history, 12-lead electrocardiogram (ECG), and blood hematology and biochemistry tests, and urinalysis carried out within 3 weeks before study drug is administered. Normal renal function
* Age-related normotensive at screening, with supine (5 minutes) blood pressure in the range of 95 to 160 mmHg systolic, inclusive, and 55 to 95 mmHg diastolic, inclusive, at screening and before study drug administration
* Demographically comparable to the groups with renal impairment with respect to age (±10 years), weight (±20%), gender, and ethnicity
* Patients with impaired renal function: Has a CrCl of <80 mL/min
* Severity of renal disease has to be stable: No significant change in renal function as evidenced by the serum creatinine value within ±20% from the last determination, obtained within at least 2 months before study entry
* Is on stable dose of medication and/or treatment regimen for renal impairment from 2 months before the study. Patients with stable cardiovascular disease including hypertension controlled with a stable dose of medication for at least 2 months before enrollment, provided that the investigator feels their condition will not interfere with the results of the study. Patients with abnormal ECG changes considered by the investigator to be insignificant or clinically compatible with the patients's renal impairment may be included
* Patients on a stable dose of thyroid hormone replacement therapy, for at least 3 months before enrollment, may be enrolled, provided that the patients' condition will not interfere with the results of the study
* Patients with mild, stable, chronic degenerative joint disease may be enrolled
* Patients on concomitant medications to treat underlying disease states or medical conditions related to renal insufficiency may be enrolled into the study, except when specifically excluded by name or pharmacological class.

Exclusion Criteria:

* Patients with normal renal function: Has any significant history or presence of hematologic, gastrointestinal, renal, hepatic, cardiovascular, pulmonary, metabolic, neurologic, or psychiatric disease, has a relevant history of drug allergy, has a history of congenital or hereditary kidney disease (including polycystic kidney disease), has a history of nephrectomy
* Used any prescription or nonprescription medication (herbal supplements included) within 21 days before administration of study drug except for paracetamol (acetaminophen), hormonal contraceptives, and replacement therapy
* Patients with impaired renal function:Is in end stage renal disease, requiring dialysis, has an acute unstable and/or significant and untreated medical illness (e.g., infection, unstable angina), has any abnormality in medical history, physical examination, ECG, or laboratory results that, in the opinion of the investigator, may affect the safety of the patient (e.g., myocardial infarction, conduction defects [e.g., QTc interval >450 msec for men, >470 msec for women], atrial or ventricular arrhythmia, coronary artery disease, congestive heart failure, valvular diseases, peripheral vascular disorders, stroke, hematologic, pulmonary, neurologic, hepatic, psychiatric, metabolic or endocrine disturbances, or inadequate nutritional status, has a history of uric acid stone disease (in the last 5 years with recurrences), uricosuria, or current hyperuricemia serum uric acid >=10 mg/dL, has uncontrolled Type 1 or 2 diabetes, has or had a renal transplant, systemic lupus erythematosus, or renal carcinoma, or has moderate to severe uncontrolled hypertension, defined as DBP >=105 mmHg and/or SBP >=180 mmHg (patients with stable mild hypertension controlled by a constant regimen over the last 2 months may be enrolled).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-04; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of a single oral dose of 3 mg ER OROS paliperidone in patients with varying degrees of renal impairment (mild, moderate, and severe), compared with patients with normal renal function

SECONDARY OUTCOMES:
To assess the disposition of the (+) and (-) enantiomers, to determine plasma protein binding of the enantiomers, and to evaluate the tolerability and safety profile of ER OROS paliperidone in patients with renal impairment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the pharmacokinetics of ER OROS paliperidone in volunteers with normal or impaired renal function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=567&filename=CR004207_CSR.pdf